CLINICAL TRIAL: NCT00520676
Title: A Randomized Phase 3 Study Comparing Pemetrexed-Carboplatin With Docetaxel-Carboplatin as First-Line Treatment for Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: Chemotherapy in Treating Patients With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly and Company
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11626; H3E-CR-S380 (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-08-22; First posted 2007-08-24 (Estimated); Results first posted 2011-07-18 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2011-08

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Docetaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- pemetrexed plus carboplatin (Experimental): Drug: pemetrexed 500 milligrams per square meter (mg/m^2), intravenous (IV), every (q) 21 days x 6 cycles maximum
  Drug: carboplatin Area Under the Curve (AUC) 5 milligram*minute/milliLiter (mg*min/mL), IV, q 21 days x 6 cycles maximum
  Interventions: Drug: pemetrexed; Drug: carboplatin
- docetaxel plus carboplatin (Active Comparator): Drug: docetaxel 75 mg/m^2, IV, q 21 days x 6 cycles maximum
  Drug: carboplatin AUC 5 mg*min/mL, IV, q 21 days x 6 cycles maximum
  Interventions: Drug: docetaxel; Drug: carboplatin

INTERVENTIONS:
Drug: pemetrexed — 500 mg/m^2, IV, q 21 days x 6 cycles maximum
  Other Names: LY231514; Alimta
  Arms: pemetrexed plus carboplatin
Drug: docetaxel — 75 mg/m^2, IV, q 21 days x 6 cycles maximum
  Arms: docetaxel plus carboplatin
Drug: carboplatin — AUC 5 mg*min/mL, IV, q 21 days x 6 cycles maximum

SUMMARY:
The purpose of this study is to compare the combination of pemetrexed and carboplatin with the combination of docetaxel and carboplatin in terms of survival without Grade 3 or 4 toxicity in previously untreated patients with locally advanced or metastatic non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Patient with locally advanced or metastatic (Stage IIIB/IV) NCSLC with no prior chemotherapy for advanced disease or molecular target treatment
* Easter Cooperative Oncology Group (ECOG) performance status 0 to 2
* Estimated life expectancy of at least 8 weeks

Exclusion Criteria:

* Known or suspected brain metastases
* Concurrent administration of any other tumor therapy
* Serious concomitant disorders
* Pregnancy or breast feeding
* Inability or unwillingness to take folic acid or vitamin B12 supplementation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2007-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (20):
- Australia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ballarat, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankston, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wendouree, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bunbury, Western Australia
- Brazil (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barretos
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goiânia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santo André
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- China (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nanjing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai
- Mexico (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ciudad Obregón
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durango
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexicali
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
- South Korea (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suwon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ulsan
- Taiwan (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taoyuan District

REFERENCES:
- [Derived] Loureiro H, Kolben TM, Kiermaier A, Ruttinger D, Ahmidi N, Becker T, Bauer-Mehren A. Correlation Between Early Trends of a Prognostic Biomarker and Overall Survival in Non-Small-Cell Lung Cancer Clinical Trials. JCO Clin Cancer Inform. 2023 Sep;7:e2300062. doi: 10.1200/CCI.23.00062. PMID 37922432
- [Derived] Pereira JR, Cheng R, Orlando M, Kim JH, Barraclough H. Elderly subset analysis of randomized phase III study comparing pemetrexed plus carboplatin with docetaxel plus carboplatin as first-line treatment for patients with locally advanced or metastatic non-small cell lung cancer. Drugs R D. 2013 Dec;13(4):289-96. doi: 10.1007/s40268-013-0032-6. PMID 24277116
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Analyses were conducted on the qualified intent-to-treat population (Q-ITT) unless otherwise specified. This population includes all data from all randomized participants, with nonsquamous histology, receiving at least 1 dose of the study drug according to the treatment the participants were assigned.
Groups:
- Pemetrexed Plus Carboplatin: pemetrexed 500 mg/m^2 plus carboplatin AUC 5 mg*min/mL on Day 1 every 21 days
- Docetaxel Plus Carboplatin: docetaxel 75 mg/m^2 plus carboplatin AUC 5 mg*min/mL on Day 1 every 21 days
Period: Overall Study
Arm/Group | Pemetrexed Plus Carboplatin | Docetaxel Plus Carboplatin
Started | 128 | 132
Received at Least 1 Dose of Study Drug | 118 | 127
Qualified Intent-to-treat (Q-ITT) | 106 | 105
Completed | 27 | 29
Not Completed | 101 | 103
Not completed — Death | 84 | 81
Not completed — Lost to Follow-up | 6 | 10
Not completed — Physician Decision | 4 | 1
Not completed — Withdrawal by Subject | 7 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pemetrexed Plus Carboplatin | Docetaxel Plus Carboplatin | Total
Number analyzed (Participants) | 106 | 105 | 211
Age Continuous [Mean (Standard Deviation); unit: years] | 59.6 (10.0) | 59.2 (10.7) | 59.4 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 55 | 97
  Male | 64 | 50 | 114
Region of Enrollment [Number; unit: participants]
  Taiwan | 3 | 9 | 12
  Mexico | 17 | 22 | 39
  Brazil | 35 | 25 | 60
  Australia | 10 | 14 | 24
  China | 20 | 17 | 37
  Korea, Republic of | 21 | 18 | 39
Smoking Status [Number; unit: participants]
  Never Smoking | 34 | 41 | 75
  Ever Smoking but Quit | 61 | 53 | 114
  Currently Smoking | 11 | 11 | 22
Histology [Number; unit: participants]
  Adenocarcinoma, lung | 10 | 11 | 21
  Adenocarcinoma, not otherwise specified | 80 | 80 | 160
  Large cell carcinoma, lung | 10 | 9 | 19
  Carcinoma, lung | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Survival Without Grade 3 or 4 Toxicity
Description: Defined as the time from date of randomization to first date of a Grade 3 or 4 treatment-emergent adverse event (TEAE; as graded by the National Cancer Institute Common Terminology Criteria for Adverse Events [CTCAE], version 3.0) or death due to any cause. Grade 3 TEAE: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated. Grade 4 TEAE: Life-threatening consequences; urgent intervention indicated.
  Participants who were alive without experiencing Grade 3 or 4 toxicity were censored at the date of last contact.
Time Frame: Baseline to until 218 events (defined as death or Grade 3 or 4 toxicity) have been observed (up to 33.3 months).
Population: Analysis was performed on protocol-qualified, intent-to-treat (Q-ITT) population. This population includes all data from all randomized participants, with nonsquamous histology, receiving at least 1 dose of the study drug according to the treatment the participants were assigned.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed Plus Carboplatin | Docetaxel Plus Carboplatin
Number analyzed (Participants) | 106 | 105
months | 3.2 [2.1 to 3.7] | 0.7 [0.5 to 1.2]
Statistical Analysis 1: Comparison: Pemetrexed Plus Carboplatin vs Docetaxel Plus Carboplatin; Test type: Superiority or Other; p < 0.001, Log Rank — The comparison was conducted at a 1-sided significance level of 0.05; Note that the 2-sided p-value for log rank is reported, which is <0.001, hence 1-sided p-value is <0.001; Hazard Ratio (HR) = 0.45, 95% CI 2-sided [0.34 to 0.60] — Cox regression model is used for HR estimate

2. Secondary Outcome: Overall Survival (OS)
Description: OS is the duration from enrollment to death. For participants who are alive, OS is censored at the last contact.
Time Frame: Baseline to until 218 events (defined as death or Grade 3 or 4 toxicity) have been observed (up to 33.3 months).
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed Plus Carboplatin | Docetaxel Plus Carboplatin
Number analyzed (Participants) | 106 | 105
months | 14.9 [12.2 to 19.0] | 14.7 [10.8 to 19.8]
Statistical Analysis 1: Comparison: Pemetrexed Plus Carboplatin vs Docetaxel Plus Carboplatin; Test type: Superiority or Other; p = 0.934, Log Rank — The comparison was conducted at a 2-sided significance level of 0.05; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.72 to 1.42] — Cox regression model is used for hazard ratio (HR) estimate

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Defined as the time from date of first dose to the first observation of disease progression (PD), or death due to any cause.
Time Frame: Baseline to until 218 events (defined as death or Grade 3 or 4 toxicity) have been observed (up to 33.3 months).
Population: Analysis was performed on protocol-qualified, intent-to-treat (Q-ITT) population. This set includes all data from all randomized participants, with nonsquamous histology, receiving at least 1 dose of the study drug according to the treatment the participants were assigned.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed Plus Carboplatin | Docetaxel Plus Carboplatin
Number analyzed (Participants) | 106 | 105
months | 5.8 [4.8 to 6.4] | 6.0 [4.8 to 6.6]
Statistical Analysis 1: Comparison: Pemetrexed Plus Carboplatin vs Docetaxel Plus Carboplatin; Test type: Superiority or Other; p = 0.800, Log Rank — The comparison was conducted at a 2-sided significance level of 0.05; Cox regression model is used for hazard ratio (HR) estimate; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.72 to 1.29]

4. Secondary Outcome: Percentage of Participants With Tumor Response (Response Rate)
Description: Response using Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Complete Response (CR)=disappearance of all target lesions; Partial Response (PR)=at least a 30% decrease in sum of longest diameter of target lesions; Progressive Disease (PD)=at least a 20% increase in sum of longest diameter of target lesions; Stable Disease (SD)=small changes not meeting above criteria. Response rate (%)=Number of participants with CR+PR/Number of participants analyzed *100. Disease Control rate=Number of participants with SD+PR+CR/Number of participants analyzed *100.
Time Frame: Baseline to until 218 events (defined as death or Grade 3 or 4 toxicity) have been observed (up to 33.3 months).
Population: Analysis was performed on tumour response-qualified population. This population includes all participants with locally advanced or metastatic non-small cell lung cancer (NSCLC), non-squamous histology with measurable disease as defined by RECIST (Version 1.0), who received at least 1 dose of pemetrexed, docetaxel, or carboplatin.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed Plus Carboplatin | Docetaxel Plus Carboplatin
Number analyzed (Participants) | 106 | 104
percentage of participants
  Tumor Response Rate | 34.0 [25.0 to 43.8] | 23.1 [15.4 to 32.4]
  Disease Control Rate | 74.5 [65.1 to 82.5] | 64.4 [54.4 to 73.6]
  Complete Response | 0.9 [0.0 to 5.1] | 0 [0 to 3.5]
  Partial Response | 33.0 [24.2 to 42.8] | 23.1 [15.4 to 32.4]
  Stable Disease | 40.6 [31.1 to 50.5] | 41.3 [31.8 to 51.4]
  Progressive Disease | 16.0 [9.6 to 24.4] | 17.3 [10.6 to 26.0]
  Unknown | 9.4 [4.6 to 16.7] | 18.3 [11.4 to 27.1]
Statistical Analysis 1: Comparison: Pemetrexed Plus Carboplatin vs Docetaxel Plus Carboplatin; Test type: Superiority or Other; p = 0.081, Fisher Exact — The comparison of tumor response rates was conducted at a 2-sided significance level of 0.05; Tumor response rate= # participants with a confirmed best response of CR or PR / # of participants who qualify for the analysis population; Odds Ratio (OR) = 1.71, 95% CI 2-sided [0.93 to 3.15] — Logistic regression model is used for odds ratio (OR) estimate

5. Other Pre Specified Outcome: Duration of Response
Description: The duration of a complete response (CR) or partial response (PR) was defined as the time from first objective status assessment of CR or PR to the first time of progression or death as a result of any cause. Response using Response Evaluation Criteria In Solid Tumors (RECIST) criteria. CR=disappearance of all target lesions; PR=at least a 30% decrease in sum of longest diameter of target lesions.
Time Frame: Baseline to until 218 events (defined as death or Grade 3 or 4 toxicity) have been observed (up to 33.3 months).
Population: Analysis was performed on tumour response qualified population. This population includes all participants with locally advanced or metastatic non-small cell lung cancer (NSCLC), non-squamous histology with measurable disease as defined by RECIST (Version 1.0), who received at least 1 dose of pemetrexed, docetaxel, or carboplatin.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed Plus Carboplatin | Docetaxel Plus Carboplatin
Number analyzed (Participants) | 106 | 104
months | 5.5 [4.0 to 8.1] | 5.4 [4.4 to 6.7]
Statistical Analysis 1: Comparison: Pemetrexed Plus Carboplatin vs Docetaxel Plus Carboplatin; Test type: Superiority or Other; p = 0.641, Log Rank — The comparison was conducted at a 2-sided significance level of 0.05; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.49 to 1.55] — Cox regression model is used for hazard ratio (HR) estimate

6. Secondary Outcome: Survival Without Clinically Important Grade 3 or 4 Toxicity
Description: Survival without Grade 3 or 4 toxicity is the time from date of randomization to the first date of the following clinically important Grade 3 or 4 TEAEs graded by the Common Terminology Criteria for Adverse Events [CTCAE], version 3.0: neutropenia (lasting >5 days), febrile neutropenia, documented infections related to neutropenia, anemia, thrombocytopenia, fatigue, nausea, vomiting, diarrhea, stomatitis, and neurosensory events; or death due to any cause. Participants who were alive without experiencing Grade 3 or 4 toxicity were censored for this analysis at the date of last contact.
Time Frame: Baseline to until 218 events (defined as death or Grade 3 or 4 toxicity) have been observed (up to 33.3 months).
Population: Analysis was performed on protocol-qualified, intent-to-treat (Q-ITT) population. This population includes all data from all randomized participants, with nonsquamous histology, receiving at least one dose of the study drug according to the treatment the participants were assigned.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed Plus Carboplatin | Docetaxel Plus Carboplatin
Number analyzed (Participants) | 106 | 105
months | 3.6 [3.0 to 8.0] | 1.3 [1.1 to 1.9]
Statistical Analysis 1: Comparison: Pemetrexed Plus Carboplatin vs Docetaxel Plus Carboplatin; Test type: Superiority or Other; p < 0.001, Log Rank — The comparison was conducted at a 2-sided significance level of 0.05; Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.40 to 0.71] — Cox regression model is used for unadjusted hazard ratio (HR) estimate

7. Secondary Outcome: Survival Without Grade 4 Toxicity
Description: Survival without Grade 4 toxicity is the time from the date of randomization to the first date of a Grade 4 TEAE or death due to any cause. Participants who are alive without experiencing Grade 4 toxicity will be censored for this analysis at the date of last contact.
Time Frame: Baseline to until 218 events (defined as death or Grade 4 toxicity) have been observed (up to 33.3 months).
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: participants
Arm/Group | Pemetrexed Plus Carboplatin | Docetaxel Plus Carboplatin
Number analyzed (Participants) | 106 | 105
participants | 12.2 [8.4 to 14.9] | 2.0 [1.6 to 3.8]
Statistical Analysis 1: Comparison: Pemetrexed Plus Carboplatin vs Docetaxel Plus Carboplatin; Test type: Superiority or Other; p < 0.001, Log Rank — The comparison was conducted at a 2-sided significance level of 0.05; Hazard Ratio (HR) = 0.49, 95% CI 2-sided [0.35 to 0.66] — Cox regression model is used for unadjusted hazard ratio (HR) estimate

8. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Summaries of serious AEs (SAEs) and all other non-serious AEs are located in the Reported Adverse Event Module.
Time Frame: Baseline to until 218 events (defined as death or Grade 3 or 4 toxicity) have been observed (up to 33.3 months).
Population: Analysis was performed on safety population. This population includes all participants with non-squamous histology who received at least one dose of study drug. Participants were analysed according to treatments they actually received.
Measure: Number; unit: participants
Arm/Group | Pemetrexed Plus Carboplatin | Docetaxel Plus Carboplatin
Number analyzed (Participants) | 106 | 105
participants
  Non-Serious Adverse Events (AEs) | 94 | 100
  Serious Adverse Events (SAEs) | 28 | 35

ADVERSE EVENTS:
Arm/Group | Pemetrexed Plus Carboplatin | Docetaxel Plus Carboplatin
Serious Adverse Events (participants affected / at risk) | 28/106 | 35/105
Other Adverse Events (participants affected / at risk) | 94/106 | 100/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed Plus Carboplatin (N=106) | Docetaxel Plus Carboplatin (N=105)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 9 (10)
Haematotoxicity (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 8 (9)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 3 (3)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cor pulmonale (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Asthenia (General disorders) | 1 (1) | 2 (2)
Chest pain (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 7 (7)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Body temperature increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Superior vena caval occlusion (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed Plus Carboplatin (N=106) | Docetaxel Plus Carboplatin (N=105)
Anaemia (Blood and lymphatic system disorders) | 36 (46) | 18 (25)
Leukopenia (Blood and lymphatic system disorders) | 33 (80) | 56 (139)
Lymphopenia (Blood and lymphatic system disorders) | 14 (26) | 25 (38)
Neutropenia (Blood and lymphatic system disorders) | 40 (109) | 74 (203)
Thrombocytopenia (Blood and lymphatic system disorders) | 12 (23) | 4 (6)
Arrhythmia (Cardiac disorders) | 3 (3) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 11 (14) | 13 (16)
Constipation (Gastrointestinal disorders) | 18 (23) | 15 (17)
Diarrhoea (Gastrointestinal disorders) | 12 (21) | 30 (43)
Dyspepsia (Gastrointestinal disorders) | 5 (6) | 7 (8)
Nausea (Gastrointestinal disorders) | 43 (71) | 37 (66)
Stomatitis (Gastrointestinal disorders) | 9 (17) | 11 (16)
Vomiting (Gastrointestinal disorders) | 18 (22) | 19 (31)
Asthenia (General disorders) | 15 (20) | 19 (30)
Chest pain (General disorders) | 4 (4) | 7 (7)
Fatigue (General disorders) | 13 (15) | 21 (24)
Mucosal inflammation (General disorders) | 7 (11) | 5 (7)
Oedema (General disorders) | 4 (4) | 6 (6)
Pyrexia (General disorders) | 11 (12) | 7 (15)
Conjunctivitis infective (Infections and infestations) | 7 (8) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 7 (7)
Alanine aminotransferase increased (Investigations) | 9 (11) | 3 (3)
Platelet count decreased (Investigations) | 7 (13) | 5 (11)
Weight decreased (Investigations) | 3 (3) | 6 (6)
Decreased appetite (Metabolism and nutrition disorders) | 27 (37) | 30 (35)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 8 (11)
Dizziness (Nervous system disorders) | 7 (8) | 7 (7)
Dysgeusia (Nervous system disorders) | 7 (12) | 11 (15)
Headache (Nervous system disorders) | 8 (9) | 7 (9)
Neurotoxicity (Nervous system disorders) | 2 (2) | 7 (11)
Paraesthesia (Nervous system disorders) | 0 (0) | 7 (8)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (10) | 14 (18)
Insomnia (Psychiatric disorders) | 7 (7) | 6 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 8 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 10 (10)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 10 (11) | 45 (46)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (8) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 8 (9) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days